CLINICAL TRIAL: NCT05189262
Title: Extra-Cellular Hemoglobin, Organ Injury in Extended Cardiopulmonary Bypass
Brief Title: Cardiopulmonary Bypass Induced Red Blood Cell Lysis
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Paul Buehler, Research Faculty, University of Maryland, Baltimore
Other Study IDs: HP-00094849; 1R01HL162120-01 (NIH)
Record Dates: First submitted 2021-11-09; First posted 2022-01-12 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cardiopulmonary Bypass; Cardiac Surgery; Kidney Injury, Acute
MeSH Terms: conditions — Acute Kidney Injury | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Red blood cells, plasma and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Sugery Patients Requiring Cardiopulmonary >1hour: Patients admitted for a complex cardiac surgery, heart valve replacement and/or CABG surgery requiring CPB >1hour
  Interventions: Other: Blood and urine collection

INTERVENTIONS:
Other: Blood and urine collection — No intervention - Biological specimen collection

SUMMARY:
Studying the dynamics of red blood cell lysis, pfH, protective proteins and organ injury, limits will be set for safe levels of pfH following the use of CPB. These results will be compared to existing laboratory-based methods for determining red blood cell damage to predict CPB assist device safety. Further, results from the studies described in this proposal will help develop therapeutic strategies to benefit patients by early detection of pfH and clearance protein levels that occur during CPB.

DETAILED DESCRIPTION:
Cost estimates for brain, lung, cardiac, and kidney complications following complex cardiac surgeries that require a medical assist device to by-pass the heart and lungs (cardiopulmonary bypass, CPB) is estimated to cost $80 million per individual states in the US over a ten-year period. These extra costs represent a significant burden on the healthcare system but could be reduced by understanding how medical assist devices lead to organ injury associated with complex cardiac surgeries. The primary goals of this research are to (1) understand how hemoglobin released into plasma (pfH) from damaged red blood cells that passage through CPB contributes to organ injury. (2) Determine the amount of pfH necessary to cause organ injury. (3) Determine the concentration changes in protective proteins (called haptoglobin, hemopexin and transferrin) that remove pfH and its degradation products from the circulation. (4) Design a computer-based model that will determine the levels of pfH and protective proteins to predict the potential for organ injury. By studying the dynamics of red blood cell lysis, pfH, protective proteins and organ injury limits will be set for safe levels of pfH following the use of CPB. These results will be compared to existing laboratory-based methods for determining red blood cell damage to predict CPB assist device safety. Further, results from the studies described in this proposal will help develop therapeutic strategies to benefit patients by early detection of pfH and clearance protein levels that occur during CPB. The primary goals of this research are to (1) understand how hemoglobin released into plasma (pfH) from damaged red blood cells that passage through CPB contributes to organ injury. (2) Determine the amount of pfH necessary to cause organ injury. (3) Determine the concentration changes in protective proteins (called haptoglobin, hemopexin and transferrin) that remove pfH and its degradation products from the circulation. (4) Design a computer-based model that will determine the levels of pfH and protective proteins to predict the potential for organ injury. By studying the dynamics of red blood cell lysis, pfH, protective proteins and organ injury limits will be set for safe levels of pfH following the use of CPB. These results will be compared to existing laboratory-based methods for determining red blood cell damage to predict CPB assist device safety. Further, results from the studies described in this proposal will help develop therapeutic strategies to benefit patients by early detection of pfH and clearance protein levels that occur during CPB.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to UMMC for cardiac procedure
* Age: >/=18 y.o TO 88 y.o.
* Undergoing CPB >1hr for the following surgeries (a) complex cardiac surgery (b) heart valve replacement surgery OR (c) CABG surgery.

Exclusion Criteria:

* Pregnant
* Non English speaking
* Unable to consent or have Legally Authorized Representative (LAR) assent to study

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Research Participants will include approximately 90 adult (>/=18 years of age to 75 years of age) medium to high risk patients. Both Male and female subjects who are undergoing complex cardiac surgery requiring, heart valve replacement, or CABG surgery requiring cardiopulmonary bypass >1hr will be eligible for enrollment at the University of Maryland Medical Center (UMMC) in Baltimore, MD. This study is a prospective observational investigation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Hemolysis | Change from baseline at hour 1 during procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron
Hemolysis | Change from baseline at hour 2 during procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron
Hemolysis | Change from baseline at hour 3 during procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron
Hemolysis | Change from baseline at hour 4 during procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron etc.
  Change from Baseline at Hour 1 during procedure
Hemolysis | Change from baseline at hour 4 post procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron etc.
  Change from Baseline at Hour 1 during procedure
Hemolysis | Change from baseline at hour 2 post procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron etc.
  Change from Baseline at Hour 1 during procedure
Hemolysis | Change from baseline at hour 24 post procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron etc.
  Change from Baseline at Hour 1 during procedure
Hemolysis | Change from baseline on day 2 post procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron etc.
  Change from Baseline at Hour 1 during procedure
Hemolysis | Change from baseline on day 3 post procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron etc.
  Change from Baseline at Hour 1 during procedure
Hemolysis | Change from baseline on day 4 post procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron etc.
  Change from Baseline at Hour 1 during procedure
Hemolysis | Change from baseline on day 5 post procedure
  Change in Measure hemoglobin released into plasma (pfH), lactate dehydrogenase and iron etc.
  Change from Baseline at Hour 1 during procedure

SECONDARY OUTCOMES:
Kidney injury | Change from baseline at hour 1 during procedure
  Change in creatinine, KIM-1 and NGAL
Kidney injury | Change from baseline at hour 2 during procedure
  Change in creatinine, KIM-1 and NGAL
Kidney injury | Change from baseline at hour 3 during procedure
  Change in creatinine, KIM-1 and NGAL
Kidney injury | Change from baseline at hour 4 during procedure
  Change in creatinine, KIM-1 and NGAL
Kidney injury | Change from baseline at hour 2 post procedure
  Change in creatinine, KIM-1 and NGAL
Kidney injury | Change from baseline at hour 24 post procedure
  Change in creatinine, KIM-1 and NGAL
Kidney injury | Change from baseline at 2 days post procedure
  Change in creatinine, KIM-1 and NGAL
Kidney injury | Change from baseline at 3 days post procedure
  Change in creatinine, KIM-1 and NGAL
Kidney injury | Change from baseline at 4 days post procedure
  Change in creatinine, KIM-1 and NGAL
Kidney injury | Change from baseline at 5 days post procedure
  Change in creatinine, KIM-1 and NGAL

OTHER OUTCOMES:
Blood cell function | Change from baseline at hour 1 during procedure
  CBC and red blood cell deformability
Blood cell function | Change from baseline at hour 2 during procedure
  CBC and red blood cell deformability
Blood cell function | Change from baseline at hour 3 during procedure
  CBC and red blood cell deformability
Blood cell function | Change from baseline at hour 4 during procedure
  CBC and red blood cell deformability
Blood cell function | Change from baseline at hour 2 post procedure
  CBC and red blood cell deformability
Blood cell function | Change from baseline at hour 24 post procedure
  CBC and red blood cell deformability
Blood cell function | Change from baseline at day 2 post procedure
  CBC and red blood cell deformability
Blood cell function | Change from baseline at day 3 post procedure
  CBC and red blood cell deformability
Blood cell function | Change from baseline at day 4 post procedure
  CBC and red blood cell deformability
Blood cell function | Change from baseline at day 5 post procedure
  CBC and red blood cell deformability
Outcome Hemoglobin Clearance | Change from baseline at hour 1 during procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations
Outcome Hemoglobin Clearance | Change from baseline at hour 2 during procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations
Outcome Hemoglobin Clearance | Change from baseline at hour 3 during procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations
Outcome Hemoglobin Clearance | Change from baseline at hour 4 during procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations
Outcome Hemoglobin Clearance | Change from baseline at hour 2 post procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations
Outcome Hemoglobin Clearance | Change from baseline at hour 24 post procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations
Outcome Hemoglobin Clearance | Change from baseline at day 2 post procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations
Outcome Hemoglobin Clearance | Change from baseline at day 3 post procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations
Outcome Hemoglobin Clearance | Change from baseline at day 4 post procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations
Outcome Hemoglobin Clearance | Change from baseline at day 5 post procedure
  Change in hemoglobin clearance measured by plasma haptoglobin and transferrin concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Paul Buehler, PhD, Principal Investigator — University of Maryland
Locations (1):
- Center for Blood Oxygen Transport and Hemostasis, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data may be used in a publication